CLINICAL TRIAL: NCT06048237
Title: Reliability of Diaphragm Thickness and Excursion Measurements Performed Via Rehabilitative Ultrasound Imaging (RUSI) Across Healthy Parous and Nulliparous Women
Brief Title: Investigating Diaphragm Thickness and Mobility in Healthy Parous and Nulliparous Volunteers Using RUSI
Status: Completed | Type: Observational
Sponsor: Evdokia Billis (Other)
Collaborators: University of Crete (Other); University of Thessaly (Other)
Responsible Party: Sponsor-Investigator, Evdokia Billis, Professor in Physiotherapy, University of Patras
Organization: University of Patras (Other)
Other Study IDs: RUSI and diaphragm
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2023-12

CONDITIONS: Asymptomatic Condition
Keywords: Ultrasound; Diaphragm/diagnostic imaging; Rehabilitation; Parity; Validation Study
MeSH Terms: conditions — Asymptomatic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Reliability Assessment Arm: This is a single-arm reliability assessment study. Reliability will be assessed by conducting measurements of diaphragm thickness and excursion on the same participants by the same rater (intra-rater reliability) and by different raters (inter-rater reliability) to evaluate measurement consistency.
  Interventions: Diagnostic Test: Diagnostic Ultrasound Imaging of the diaphragm

INTERVENTIONS:
Diagnostic Test: Diagnostic Ultrasound Imaging of the diaphragm — In this reliability study, ultrasound imaging will be utilized by trained physiotherapists to assess diaphragm thickness and excursion. Participants will be positioned in a semi-recumbent position, while the scanning area will be marked with a surgical skin marker according to specific anatomical landmarks recommended, to ensure reproducibility of the procedure. Ultrasound probe will be placed at the zone of apposition to visualize the diaphragm through the liver window.
  Diaphragm thickness will be assessed during both full inhalation and exhalation, capturing images in B-mode to measure distance between the diaphragmatic pleura and peritoneal fascia. Diaphragm excursion will be assessed during tidal volume diaphragmatic breathing, using M-mode to track the craniocaudal displacement of the diaphragm during respiratory cycle. Data obtained will contribute to the evaluation of the reliability of diaphragm thickness and excursion measurements for potential future clinical applications.

SUMMARY:
The purpose of this study is to evaluate the intra-rater and inter-rater reliability of diaphragm thickness and excursion measurements by applying Rehabilitative Ultrasound Imaging (RUSI) in a diverse cohort of healthy women, including nulliparous and parous across varying age groups.

The diaphragm, which is primarily a respiratory muscle, is also considered to contribute to spinal stability. Utilizing RUSI, a non-invasive and cost-effective imaging modality, we intend to examine diaphragm parameters. Preliminary evidence highlights a potential link between diaphragm dysfunction and musculoskeletal conditions such as lumbopelvic pain. This research hypothesizes that understanding diaphragm behavior in different pathologies, including postpartum recovery and lower back pain, can contribute to tailored rehabilitation strategies, potentially benefiting a wide range of clinical conditions, and facilitating the assessment of intervention effectiveness. Additionally, this study addresses the lack of research on the diaphragm's role in postpartum rehabilitation and offers novel insights into its reliability, particularly within this demographic.

DETAILED DESCRIPTION:
The diaphragm is the main respiratory muscle but is also considered to contribute significantly to trunk stability and posture due to its unique anatomy and coordination with other trunk muscles. Rehabilitative Ultrasound Imaging (RUSI) technique provides a safe, and cost-effective method for assessing diaphragm muscle function. RUSI is employed in musculoskeletal physiotherapy to assess diaphragm thickness or mobility in trunk conditions such as lumbopelvic pain, as a method to investigate rehabilitation effectiveness or as a biofeedback tool for muscle training. Although, the reliability of RUSI measurements for diaphragm thickness and excursion has been previously investigated in healthy populations, individuals with pelvic girdle pain and athletes with lumbopelvic pain, its reliability on postpartum populations has never been researched. Therefore, this study aims to assess the reliability of diaphragm thickness and excursion measurements in healthy women, including nulliparous and parous individuals of varying ages, utilizing RUSI.

This reliability study adheres to Ethical considerations and the Helsinki Declaration and is approved by the Research Ethics Committee (R.E.C.) of the University of Patras. The study incorporates a robust quality assurance plan, according to the Internal Review Board of the Research Ethics Committee (R.E.C.) of the University of Patras, including data checks to assess data validation and registry procedures performed by the Data Monitoring Committee of R.E.C. of the University of Patras, as well as site monitoring and auditing, to maintain protocol adherence and data collection integrity. The accuracy, completeness, and representativeness of registry data is assured by the research team, comparing the data to preliminary data published in similar reliability studies. A comprehensive data dictionary is established among the research team, containing detailed variable descriptions, coding information, and normal ranges, ensuring consistency and clarity in data collection.

RUSI is performed by two trained physiotherapists (with more than 5 years of clinical experience in musculoskeletal physiotherapy). The physiotherapists received one-day training from a consultant radiologist, specializing in musculoskeletal sonographic imaging, followed by several hours of independent and joint practice between the radiologist and physiotherapists. A convenience sample of adult women coming from around the broader university campus area is invited to participate in the study, via advertisements and university-mediated means (emails, e-platform university announcements etc.). Informed consent is obtained from all participants. Participants undergo an ultrasound assessment in the semi-recumbent position with the Versana Active™ ultrasound system. Anatomical guide points are marked by a surgical skin marker for accuracy, and the 2 trained physiotherapists perform the assessments according to Boussuges et al. (2020) recommendations. Diaphragm thickness is measured using a high-resolution linear transducer in B-mode at the end of a full inspiration and full expiration. Diaphragm excursion is assessed using a high-resolution curvilinear transducer in M-mode during tidal volume diaphragmatic breathing. A two-minute resting interval follows each measurement. During the resting intervals, calipers are placed on the captured images according to literature recommendations and measurements are recorded and saved. Intra-tester and inter-tester reliability are evaluated by taking 3 consecutive measurements per parameter. Operators and subjects are blinded for all measurements taken, by covering measurement tables at the edge of the ultrasound screen. An independent researcher blinded to the subject identity (the identity of the subject on the ultrasound screen is concealed by the operator at the end of the assessment) and the examination procedure is responsible for the extraction, and documentation of all variables in a spreadsheet software.

All patient data are stored anonymously/coded in a secure cloud platform accessed only by the research team members. Imputation methods will be applied to address situations where variables are missing, uninterpretable, or inconsistent. Any adverse events will be addressed and documented, while medical consultation will be accessible during patient assessment hours. Any modifications to the study protocol, data collection methods, or other aspects of the study will be reviewed thoroughly among researchers and the Internal Review Board of the R.E.C., and the study protocol as well as study registration will be adjusted accordingly. Statistical analysis of the data will be performed using SPSS software (version 28.0; SPSS Inc, Chicago, IL). Reliability will be calculated using intraclass correlation coefficient (ICC) assessed with a two-way random effect model (ICC2,1) and 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy women
* Nulliparous and parous individuals
* Age between 18 and 60 years

Exclusion Criteria:

* Severe chronic respiratory conditions (e.g., COPD, chronic bronchitis, pulmonary emphysema or fibrosis)
* Body mass index (BMI) greater than 30 kg/m², which may hinder ultrasound imaging
* History of major abdominal surgery
* Pregnancy
* Neuromuscular disorders that could alter diaphragm morphology and function

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study aims to investigate the reliability of ultrasound measurements for assessing diaphragm thickness and excursion in a diverse group of healthy women, including nulliparous and parous. Being part of a bigger project protocol, there has been a lack of research into the diaphragm's stabilizing role in this specific population, and diaphragm thickness and mobility in postpartum individuals has never been investigated. Therefore, the study's secondary objective is to bridge these gaps in the existing literature by including both parous and nulliparous women in the sample. This approach seeks to provide more precise insights into the diaphragm's function as a stabilizer during the postpartum period and to compare its behavior with that of nulliparous women.
Study Population: The population from which the cohort will be selected consists of generally healthy women aged 18 to 60 years affiliated with the university campus area (professors and students from all academic levels). This population will be invited to participate through advertisements and university-mediated means, including emails and e-platform announcements.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Inspiratory Diaphragm Thickness | Measured at full inspiration during the same session (aprox. 10 minutes)
  The thickness of the diaphragm muscle at the end of a full inspiration measured in centimeters (cm).
Expiratory Diaphragm Thickness | Measured at full expiration during the same session (aprox. 10 minutes)
  The thickness of the diaphragm muscle at the end of a full expiration measured in centimeters (cm).
Diaphragm Excursion | Measured during quiet, tidal breathing during the same session in a random order (before or after diaphragm thickness) (aprox. 10 minutes)
  It measures the craniocaudal displacement (movement from top to bottom) of the diaphragm during the respiratory cycle in centimeters (cm).

SECONDARY OUTCOMES:
Thickening Fraction (Percentage of Thickening) | Thickening fraction is calculated post-assessment by an independent researcher (aprox. 5 minutes)
  This metric quantifies the percentage of change in diaphragm thickness during breathing. It is computed by taking the difference between diaphragm thickness at the end of inspiration and diaphragm thickness at the end of expiration, divided by diaphragm thickness at the end of expiration, and then multiplying by 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Billis, PhD, Study Director — University of Patras
Locations (1):
- Laboratory of Clinical Physiotherapy and Research (CPRlab), Pátrai, Achaia, Greece

IPD SHARING:
Plan to Share IPD: No
We are happy to share data if needed.

REFERENCES:
- [Background] Hodges PW, Butler JE, McKenzie DK, Gandevia SC. Contraction of the human diaphragm during rapid postural adjustments. J Physiol. 1997 Dec 1;505 ( Pt 2)(Pt 2):539-48. doi: 10.1111/j.1469-7793.1997.539bb.x. PMID 9423192
- [Background] Hodges PW, Gandevia SC. Activation of the human diaphragm during a repetitive postural task. J Physiol. 2000 Jan 1;522 Pt 1(Pt 1):165-75. doi: 10.1111/j.1469-7793.2000.t01-1-00165.xm. PMID 10618161
- [Background] Shirley D, Hodges PW, Eriksson AE, Gandevia SC. Spinal stiffness changes throughout the respiratory cycle. J Appl Physiol (1985). 2003 Oct;95(4):1467-75. doi: 10.1152/japplphysiol.00939.2002. PMID 12970374
- [Background] Hodges PW, Eriksson AE, Shirley D, Gandevia SC. Intra-abdominal pressure increases stiffness of the lumbar spine. J Biomech. 2005 Sep;38(9):1873-80. doi: 10.1016/j.jbiomech.2004.08.016. PMID 16023475
- [Background] Janssens L, McConnell AK, Pijnenburg M, Claeys K, Goossens N, Lysens R, Troosters T, Brumagne S. Inspiratory muscle training affects proprioceptive use and low back pain. Med Sci Sports Exerc. 2015 Jan;47(1):12-9. doi: 10.1249/MSS.0000000000000385. PMID 24870567
- [Background] Dulger E, Bilgin S, Bulut E, Inal Ince D, Kose N, Turkmen C, Cetin H, Karakaya J. The effect of stabilization exercises on diaphragm muscle thickness and movement in women with low back pain. J Back Musculoskelet Rehabil. 2018;31(2):323-329. doi: 10.3233/BMR-169749. PMID 29278870
- [Background] Calvo-Lobo C, Almazan-Polo J, Becerro-de-Bengoa-Vallejo R, Losa-Iglesias ME, Palomo-Lopez P, Rodriguez-Sanz D, Lopez-Lopez D. Ultrasonography comparison of diaphragm thickness and excursion between athletes with and without lumbopelvic pain. Phys Ther Sport. 2019 May;37:128-137. doi: 10.1016/j.ptsp.2019.03.015. Epub 2019 Mar 28. PMID 30954705
- [Background] Scarlata S, Mancini D, Laudisio A, Benigni A, Antonelli Incalzi R. Reproducibility and Clinical Correlates of Supine Diaphragmatic Motion Measured by M-Mode Ultrasonography in Healthy Volunteers. Respiration. 2018;96(3):259-266. doi: 10.1159/000489229. Epub 2018 Aug 16. PMID 30114702
- [Background] Scarlata S, Mancini D, Laudisio A, Raffaele AI. Reproducibility of diaphragmatic thickness measured by M-mode ultrasonography in healthy volunteers. Respir Physiol Neurobiol. 2019 Feb;260:58-62. doi: 10.1016/j.resp.2018.12.004. Epub 2018 Dec 13. PMID 30553945
- [Background] Wilches-Luna EC, Pabon-Munoz FE, Arias-Campo JM, Caballero-Lozada AF. Inter-rater reliability of the measurement of diaphragmatic excursion and fraction of diaphragmatic thickening by ultrasonography in healthy volunteers. Rev Esp Anestesiol Reanim (Engl Ed). 2022 Nov;69(9):536-543. doi: 10.1016/j.redare.2021.06.003. Epub 2022 Oct 11. PMID 36241512
- [Background] Boussuges A, Rives S, Finance J, Bregeon F. Assessment of diaphragmatic function by ultrasonography: Current approach and perspectives. World J Clin Cases. 2020 Jun 26;8(12):2408-2424. doi: 10.12998/wjcc.v8.i12.2408. PMID 32607319